CLINICAL TRIAL: NCT00743457
Title: Pediatric Ocular Ultrasound for VPS Failure
Brief Title: Study of Ultrasound of the Eye for Children With Suspected Shunt Failure
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Garth Meckler, Associate Professor, Oregon Health and Science University
Other Study IDs: IRB00004484
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Hydrocephalus
Keywords: Possible VPS failure with symptom such as headache; vomiting; lethargy; VPS failure
MeSH Terms: conditions — Hydrocephalus; Vomiting; Lethargy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VPS Patients: Children 6 months-18 years with VPS and symptoms of possible shunt failure
  Interventions: Device: Ocular Ultrasound

INTERVENTIONS:
Device: Ocular Ultrasound — B-mode ultrasound of the eye with 90 and 30 degree view of optic nerve sheath

SUMMARY:
The purpose of the study is to determine whether an ultrasound of the eye can be used as a radiation-free alternative to X-ray to identify children with risk of shunt failure in the Emergency Department. Please note that a shunt is an artificial or natural channel running between two other channels.2. Briefly summarize how participants are recruited.

DETAILED DESCRIPTION:
Children (6 months to 18 years old) with ventriculoperitoneal shunts presenting to the Emergency Department (ED) with signs and symptoms of shunt failure will be recruited through their parent/legal guardian when the parent/guardian brings the child to the emergency room. Ventriculoperitoneal shunt is a device implanted surgically to relieve pressure inside the skull (intracranial pressure) caused by water on the brain (hydrocephalus).

Screening for the study includes a check of the child's age and the diagnosis by CRISP volunteer research assistants in the ED between 08:00 and 23:00. If the child is eligible, the CRISP volunteer research assistants will contact the study team. Parents/guardians will be informed by the study team of the availability of the study and will be asked if they would like to have the study explained to them and if they would like to read the consent form regarding the study. In addition to that, assent of children over 7 years of age will be obtained.

Information will be collected from the child's medical record, including medical history and current and prior symptoms and illnesses. The parent/guardian will also be asked if they believe their child's illness is due to a shunt malfunction. The child will undergo a physical exam and an ultrasound of the eye where the diameter of their optic nerve (ONSD) will be recorded. The optic nerve is the nerve that carries visual messages from the retina to the brain. Standard radiographic images, obtained as part of standard of care, will be reviewed by study radiologists blinded to the ultrasound results. The study radiologist will review the radiologic imaging and record if the outcome is suggestive of shunt failure. Another study radiologist from the Casey Eye Institute will review the results of the ocular ultrasound and record if the results are optimal or not optimal. Four weeks after the child was originally taken to the emergency room, the study team will review the child's medical record for information about the child's ED diagnosis, the procedures performed during their ED visit and if the initial radiology read was suggestive of shunt failure.

The study team will complete the ED Encounter Form on the day of the child's visit to the ED. The ED Encounter Form includes one question to the parent/guardian, who will be asked if they believe their child's illness is due to a shunt malfunction.

Results will be presented using descriptive statistics. The primary outcome measure is the proportion of children with a shunt failure who are correctly identified by the ocular ultrasound and proportion of children without shunt failure who have had a negative screening test result when an ocular ultrasound is used.

ELIGIBILITY:
Inclusion Criteria:

* 6 months to 18 years with VPS
* Headache
* Vomiting
* Mental status changes

Exclusion Criteria:

* Elevated intra-ocular pressure or known globe injury

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients 6 months to 18 years of age with VPS and symptoms of potential shunt failure presenting the the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Optic Nerve Sheath Diameter | Within 4 hours of enrollment
Clinical VPS Failure | Within 4 weeks of enrollment

SECONDARY OUTCOMES:
Standard Neuro-imaging Results (CT, MRI, X-rays) | Day of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Garth D Meckler, MD, MSHS, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States